CLINICAL TRIAL: NCT05186675
Title: Efficacy and Safety of Percutaneous Superselective Adrenal Arterial Embolization in the Treatment of Primary Aldosteronism With Bilateral Idiopathic Hyperaldosteronism: A Prospective Cohort Study
Brief Title: Superselective Adrenal Arterial Embolization for Bilateral Idiopathic Hyperaldosteronism: A Prospective Cohort Study
Acronym: SAAE-BIH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021NDEFY21
Record Dates: First submitted 2021-12-25; First posted 2022-01-11 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2021-12

CONDITIONS: Primary Aldosteronism Due to Adrenal Hyperplasia (Bilateral)
Keywords: primary aldosteronism; hypertension; superselective adrenal arterial embolization
MeSH Terms: conditions — Hyperaldosteronism; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Superselective adrenal arterial embolization (Experimental): For patients with bilateral idiopathic hyperaldosteronism confirmed by adrenal venous sampling, Superselective adrenal arterial embolization（SAAE）shall be given according to the patient's wishes. The blood pressure, plasma aldosterone and potassium levels, and adverse events were assessed after SAAE. The primary endpoint was the change in home blood pressure at one months, compared with baseline.
  Interventions: Procedure: superselective adrenal arterial embolization

INTERVENTIONS:
Procedure: superselective adrenal arterial embolization — Superselective adrenal arterial embolization is an operation to inject embolic agent into adrenal artery through catheter to embolize part of adrenal gland, so as to reduce the secretion of adrenal hormone and reduce blood pressure

SUMMARY:
The most common two subtypes of primary aldosteronism (PA ) are aldosterone producing adenoma (APA) and bilateral idiopathic hyperaldosteronism (IHA). Mineralocorticoid receptor (MR) antagonists is the main treatment for bilateral IHA, because of its side effects, the treatment compliance of those patients is poor. Hence, an alternative therapy is needed in such cases. We hypothesized that superselective adrenal artery embolization (SAAE) could be a suitable alternative approach. To our knowledge, SAAE has so far not been applied to treat bilateral IHA. This study aimed to evaluate the efficacy and safety of SAAE in the treatment of PA patients with bilateral IHA.

DETAILED DESCRIPTION:
Primary aldosteronism (PA) is the most common form of secondary hypertension, accounting for more than 5% of the general hypertensive cases and 17-20% of resistant hypertension.The most common PA subtype is bilateral idiopathic hyperaldosteronism (IHA), and medical therapy with mineralocorticoid receptor antagonists (MRAs) is recommended for these patients.The clinical studies showed that PA patients had more cardiovascular events than patients with essential hypertension independent of blood pressure, and PA patients with higher plasma aldosterone levels had a higher cardiovascular risk. However, MRAs are unable to reduce the level of plasma aldosterone. Moreover, the undesirable adverse effects of MRAs also limit their wide application, particularly in men.

Superselective adrenal artery embolization (SAAE) has been used as a minimally invasive alternative for the treatment of adrenal tumors. The clinical efficacy of SAAE has been proved by a number of clinical studies. Since the efficacy and safety of SAAE was justified by the treatment of adrenal tumors and APA, we hypothesized that SAAE might cause a significant reduction of blood pressure in cases of hypertension caused by bilateral IHA. Here, we intend to conduct a prospective cohort study to demonstrate the efficacy and safety of SAAE for bilateral IHA with a one-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age 18-60 years old, regardless of gender; (2) After strict drug elution, it met the diagnostic criteria of primary aldosteronism, and bilateral idiopathic aldosteronism was confirmed by adrenal venous sampling; (3) Blood pressure conditions meet one of the following: 1) Office blood pressure ≥ 140/90mmHg; 2) Ambulatory blood pressure monitoring：whole day blood pressure > 130/80 mmHg or daytime blood pressure > 135/85 mmHg; (4) Adrenal CT showed adrenal hyperplasia, nodules or no obvious morphological abnormalities； (5) The course of hypertension is more than 6 months； (6) The patient or his legal representative shall sign the written informed consent approved by the ethics committee before screening.

Exclusion Criteria:

* (1) Primary hypertension or secondary hypertension with other causes; (2) A woman who is pregnant or lactating, or has a birth plan in the next year; (3) There are serious organic diseases, especially liver and kidney dysfunction; (4) Severe allergy to contrast medium; (5) Other serious organic diseases, life expectancy < 12 months; (6) Adrenal CT showed adenoma. (7) Patients are enrolled or want to participate in other clinical studies. During the enrollment study, the results of this study will be affected.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Ambulatory blood pressure monitoring | one month after SAAE
  24-hour ambulatory blood pressure monitor
Office blood pressure | one month after SAAE
  sphygmomanometer

SECONDARY OUTCOMES:
plasma aldosterone | one month after SAAE
  reagent
potassium levels | one month after SAAE
  reagent
adverse events | one month after SAAE
  follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Dong Yifei, Doctor, Study Director — Second Affiliated Hospital of Nanchang University
Locations (1):
- the Second Affiliated Hospital of Nanchang University, Nanchang, Jiagxi, China

IPD SHARING:
Plan to Share IPD: No
From January 2022 to December 2022, 50 cases of bilateral idiopathic aldosteronism were selected; 2023.1-2023.2 complete the follow-up of all enrolled patients; 2023.3-2023.6 statistical data, writing and publishing academic papers

REFERENCES:
- [Background] Dong H, Zou Y, He J, Deng Y, Chen Y, Song L, Xu B, Gao R, Jiang X. Superselective adrenal arterial embolization for idiopathic hyperaldosteronism: 12-month results from a proof-of-principle trial. Catheter Cardiovasc Interv. 2021 May 1;97 Suppl 2:976-981. doi: 10.1002/ccd.29554. Epub 2021 Feb 19. PMID 33605538
- [Background] Zhao Z, Liu X, Zhang H, Li Q, He H, Yan Z, Sun F, Li Y, Zhou X, Bu X, Wu H, Shen R, Zheng H, Yang G, Zhu Z; Chongqing Endocrine Hypertension Collaborative Team. Catheter-Based Adrenal Ablation Remits Primary Aldosteronism: A Randomized Medication-Controlled Trial. Circulation. 2021 Aug 17;144(7):580-582. doi: 10.1161/CIRCULATIONAHA.121.054318. Epub 2021 Aug 16. No abstract available. PMID 34398686
- [Background] Zhang H, Li Q, Liu X, Zhao Z, He H, Sun F, Hong Y, Zhou X, Li Y, Shen R, Bu X, Yan Z, Zheng H, Yang G, Zhu Z; Chongqing Endocrine Hypertension Collaborative Team. Adrenal artery ablation for primary aldosteronism without apparent aldosteronoma: An efficacy and safety, proof-of-principle trial. J Clin Hypertens (Greenwich). 2020 Sep;22(9):1618-1626. doi: 10.1111/jch.13960. Epub 2020 Aug 27. PMID 32852871
- [Background] Monticone S, Burrello J, Tizzani D, Bertello C, Viola A, Buffolo F, Gabetti L, Mengozzi G, Williams TA, Rabbia F, Veglio F, Mulatero P. Prevalence and Clinical Manifestations of Primary Aldosteronism Encountered in Primary Care Practice. J Am Coll Cardiol. 2017 Apr 11;69(14):1811-1820. doi: 10.1016/j.jacc.2017.01.052. PMID 28385310
- [Background] Funder JW, Carey RM, Mantero F, Murad MH, Reincke M, Shibata H, Stowasser M, Young WF Jr. The Management of Primary Aldosteronism: Case Detection, Diagnosis, and Treatment: An Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2016 May;101(5):1889-916. doi: 10.1210/jc.2015-4061. Epub 2016 Mar 2. PMID 26934393
- [Background] Inoue H, Nakajo M, Miyazono N, Kanetsuki I, Miyake S, Hokotate H, Iida K, Niwatsukino H, Matsumoto Y, Tanaka D, et al. Treatment of aldosteronoma with superselective intraarterial injection of absolute ethanol. Nihon Igaku Hoshasen Gakkai Zasshi. 1994 Feb 25;54(2):154-62. No abstract available. PMID 8121780
- [Background] Fowler AM, Burda JF, Kim SK. Adrenal artery embolization: anatomy, indications, and technical considerations. AJR Am J Roentgenol. 2013 Jul;201(1):190-201. doi: 10.2214/AJR.12.9507. PMID 23789675
- [Background] Inoue H, Nakajo M, Miyazono N, Nishida H, Ueno K, Hokotate H. Transcatheter arterial ablation of aldosteronomas with high-concentration ethanol: preliminary and long-term results. AJR Am J Roentgenol. 1997 May;168(5):1241-5. doi: 10.2214/ajr.168.5.9129420.
- [Background] Hokotate H, Inoue H, Baba Y, Tsuchimochi S, Nakajo M. Aldosteronomas: experience with superselective adrenal arterial embolization in 33 cases. Radiology. 2003 May;227(2):401-6. doi: 10.1148/radiol.2272011798. Epub 2003 Apr 3. PMID 12676966
- [Background] Kometani M, Yoneda T, Demura M, Karashima S, Mori S, Oe M, Sawamura T, Okuda R, Yamagishi M, Takeda Y. The Long-term Effect of Adrenal Arterial Embolization for Unilateral Primary Aldosteronism on Cardiorenovascular Protection, Blood Pressure, and the Endocrinological Profile. Intern Med. 2016;55(7):769-73. doi: 10.2169/internalmedicine.55.5196. Epub 2016 Apr 1. PMID 27041162